CLINICAL TRIAL: NCT01275300
Title: A Pilot Study to Measure Plasma and Urinary Prostaglandin D2 Metabolites Evoked by Niacin
Brief Title: Biosynthesis of PGD2 in Vivo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 806115 - FitzGerald, MD
Record Dates: First submitted 2010-12-16; First posted 2011-01-12 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Aspirin; Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo phase I (Placebo Comparator): Subjects were given 5 days of placebo. On day 5, they were given a single dose of niacin (600 mg) administered 30 minutes after the last dose of placebo. Urine was collected sequentially for analysis. The same subjects came back for cross-over study and were assigned to Aspirin group. There was a 2-week washout period between each treatment.
  Interventions: Drug: Placebo; Drug: Niacin
- Aspirin phase I (Active Comparator): Subjects were given 5 days of 81 mg aspirin. On day 5, they were given a single dose of niacin (600 mg) administered 30 minutes after the last dose of aspirin or placebo. Urine was collected sequentially for analysis.
  Interventions: Drug: Aspirin; Drug: Niacin
- Aspirin phase II (Active Comparator): In phase II study, subjects were given 5 days of 81 mg aspirin. On day 6, they were given a single dose of niacin (600 mg) administered 24 hours after the last dose of aspirin. Urine was collected sequentially for analysis
  Interventions: Drug: Aspirin; Drug: Niacin

INTERVENTIONS:
Drug: Aspirin
  Other Names: Aspirin 81 mg
  Arms: Aspirin phase I; Aspirin phase II
Drug: Placebo
  Arms: Placebo phase I
Drug: Niacin
  Other Names: Niacin 600 mg

SUMMARY:
The investigator would like to see if aspirin could block niacin-induced flushing by analyzing blood and urine after taking aspirin.

Phase I: Subjects were assigned to either placebo or aspirin groups. They were given 5 days of 81 mg aspirin or placebo. On day 5, they were given a single dose of niacin (600 mg) administered 30 minutes after the last dose of aspirin or placebo. The same subjects came back for cross-over study and were assigned to a different group. There was a 2-week washout period between each treatment. Urine was collected sequentially for analysis

Phase II: The same study subjects come back for an open label one week study. They were given 5 days of taking 81 mg Aspirin, taken once daily, followed by a single dose of 600 mg Niacin on day 6. Urine was collected sequentially for analysis

DETAILED DESCRIPTION:
The purpose of this study is to look at the roles of various blood cells and their contributions of different prostaglandins. The intention is that by better understanding these prostaglandins and various metabolites, it will provide insights into their roles in the cardiovascular system.

Prostaglandins and metabolites are naturally occurring substances found in the blood and urine which can act as markers which can be quantified and studied as we will be doing in this study. Flushing response to niacin will also be assessed by laser doppler measuring blood flow of the facial skin.

Untransformed and transformed data will be subjected to exploratory analysis of variance appropriated for a three factor design with one two period crossover factor and two non-repeated factors. Additionally, volunteer's test(s) for paired observations will characterize the magnitude of the niacin effect on the response variables within selected time points.

ELIGIBILITY:
Inclusion Criteria:

age between 18-70

* subject must be in good health as based on medical history
* All subjects must be non-smoking, non-pregnant volunteers
* Female subjects of child bearing potential must be using a medically acceptable method of contraception throughout the entire study period. All female subjects must consent to a urine pregnancy test at screening and just prior to the start of each treatment period of the study, which must be negative at all time points.

Exclusion Criteria:

* subjects with any medical condition that according to the investigator may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject.
* subjects who have received an experimental drug within 30 days prior to the study.
* subjects who have taken medications at least 10 days prior to the study. Birth Control pills are acceptable and shall not be excluded.
* Subjects who have taken aspirin or aspirin containing products for at least 10 days prior to the study.
* Subjects who have taken acetaminophen, NSAIDS, COX-2 inhibitors (OTC or prescription) for at least 10 days prior to the study.
* Subjects who are currently consuming any type of tobacco product(s).
* Subjects who consume high doses of antioxidant vitamins daily (vitamin C > 1000mg, Vitamin E > 400 IU, Beta Carotene > 1000IU, Vitamin A > 5000IU, Selenium > 200mcg, Folic Acid > 1mg) for the 2 weeks prior to the start of the study and throughout the study.
* Subjects who consume alcohol, caffeine or high fat food 24 hours prior to study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wenliang Song, MD, Principal Investigator — University of Pennsylvania; Garret FitzGerald, MD, Study Chair — University of Pennsylvania
Locations (1):
- University of Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Song WL, Stubbe J, Ricciotti E, Alamuddin N, Ibrahim S, Crichton I, Prempeh M, Lawson JA, Wilensky RL, Rasmussen LM, Pure E, FitzGerald GA. Niacin and biosynthesis of PGD(2)by platelet COX-1 in mice and humans. J Clin Invest. 2012 Apr;122(4):1459-68. doi: 10.1172/JCI59262. Epub 2012 Mar 12. PMID 22406532
- See also: Niacin and biosynthesis of PGD2 by platelet COX-1 in mice and humans — http://www.jci.org/articles/view/59262/cite

RESULTS

PARTICIPANT FLOW:
Groups:
- "Placebo+Niacin First, Then Aspirin+Niacin; Aspirin+Niacin First, Then Placebo+Niacin: Phase I: Subjects were assigned to either placebo or aspirin groups. They were given 5 days of 81 mg aspirin or placebo. On day 5, they were given a single dose of niacin (600 mg) administered 30 minutes after the last dose of aspirin or placebo. The same subjects came back for cross-over study and were assigned to a different group. There was a 2-week washout period between each treatment. Urine was collected sequentially for analysis
  Phase II: The same study subjects come back for an open label one week study. They were given 5 days of taking 81 mg Aspirin, taken once daily, followed by a single dose of 600 mg Niacin on day 6. Urine was collected sequentially for analysis
Period: 1st Intervention (5 Days)
Arm/Group | "Placebo+Niacin First, Then Aspirin+Niacin | Aspirin+Niacin First, Then Placebo+Niacin
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | "Placebo+Niacin First, Then Aspirin+Niacin | Aspirin+Niacin First, Then Placebo+Niacin
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: 2nd Intervention(5 Days)
Arm/Group | "Placebo+Niacin First, Then Aspirin+Niacin | Aspirin+Niacin First, Then Placebo+Niacin
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | "Placebo+Niacin First, Then Aspirin+Niacin | Aspirin+Niacin First, Then Placebo+Niacin
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Phase 2: Open-label 6days)
Arm/Group | "Placebo+Niacin First, Then Aspirin+Niacin | Aspirin+Niacin First, Then Placebo+Niacin
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants had the same experience of interventions throughout the study, just in different randomized orders of receipt.
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change of Area Under Curve for the Urinary Prostaglandins Concentration Versus Time Curve (AUC) in Response to Aspirin or Placebo
Description: Percentage change of area under the urinary prostaglandins concentration versus time curve (AUC) in response to niacin with or without pretreatment of aspirin was studied. This outcome measures whether aspirin instead of placebo will impact the subjects' response to niacin. The area was normalized by percentile.
Time Frame: -2-0, 0-2, 2-4, 4-6, 6-12 and 12-24 hours pre or post niacin
Measure: Mean (95% Confidence Interval); unit: Percentage change of area under curve
Arm/Group | Placebo | Aspirin
Number analyzed (Participants) | 9 | 9
Percentage change of area under curve | 95 [93 to 97] | 43 [38 to 48]

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- P1: Placebo/Aspirin Followed by Niacin: Phase 1, 5 days of placebo, followed by a single dose of 600mg niacin on day 6, 10 day washout and 5 days of aspirin 81 mg x followed by a single dose of 600 mg niacin on day 6
  P1, placebo/aspirin followed by niacin: 5 days of placebo or aspirin followed by 600 mg niacin, 10 day washout in between two 6-day study periods
- P2: Aspirin and Niacin: Phase 2, aspirin 81 mg x 5 days and a single dose of 600 mg niacin on day 6
  P2, aspirin and niacin: aspirin 81 mg x 5 days and a single dose niacin on day 6
Arm/Group | P1: Placebo/Aspirin Followed by Niacin | P2: Aspirin and Niacin
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No